CLINICAL TRIAL: NCT01197443
Title: Parents as the Agent of Change for Childhood Obesity
Acronym: PAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kerri Boutelle, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 071669
Record Dates: First submitted 2010-08-17; First posted 2010-09-09 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
Keywords: obesity; overweight; overweight children; overweight parents; families with overweight child; body mass index; BMI; weight; childhood obesity; diet; treatment; parent modeling; traffic light diet; stop light diet
MeSH Terms: conditions — Obesity; Overweight; Body Weight; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent-only Group (Experimental): Treatment will be administered to parents of the overweight child. Parent-only group treatment will include all of the same skills and techniques to promote weight loss, but the information will be delivered only to the parent. Participation of the children assigned to the parent-only treatment arm will be limited to the baseline and follow-up assessments.
  Interventions: Behavioral: Parent-only Group
- Parent + child Group (Active Comparator): The treatment for participants in the parent + child arm will be administered in two separate groups, one for the parents and one for the child.
  Interventions: Behavioral: Parent + Child Group

INTERVENTIONS:
Behavioral: Parent-only Group — Parent-only group will include the same skills and techniques to promote weight loss as given to the parent + child group, but the information will be delivered only to the parent. Parent group will be compared to the parent group of the parent + child treatment arm. The focus will be on implementing skills learned to assist the child in weight management. The treatment length is set for 12 weekly meetings and bi-monthly meetings during months 4 and 5. Each group session will be 60-min including weigh-ins. Group meetings focus on behavior change, weight loss, healthy eating and activity for the overweight child and parent.
  Other Names: Parents as the Agent of Change for Childhood Obesity (PAAC)
  Arms: Parent-only Group
Behavioral: Parent + Child Group — The treatment for participants in the parent + child group will be administered in two separate groups, one for the parents and one for the child. Treatment will include the same skills and techniques to promote weight loss as given to the parent-only group, but the information will be delivered to both the parent and child. The treatment length, session schedule, treatment content and follow-up assessments are same as the parent-only group.
  Other Names: Parents as the Agent of Change for Childhood Obesity (PAAC)
  Arms: Parent + child Group

SUMMARY:
The overall intent of this study is to explore a promising mode for delivering treatment for childhood obesity via parent education only, and to evaluate the cost effectiveness compared to the current gold standard treatment of parent-and-child dual education.

DETAILED DESCRIPTION:
This study is a randomized clinical trial in which 150 overweight 8-12 year old children and their parent will be randomly assigned by the gender of the child to one of two conditions; a parent-only intervention or a parent + child intervention. Both treatment arms will provide behavioral treatment for childhood obesity for 5 months, and participants will be followed for 18-months post-treatment. Assessments will occur at baseline, immediately post-treatment, 6-12- and 18-months post-treatment. The overall intent of this study is to explore a promising mode for delivering treatment for childhood obesity (parent-only), and to evaluate the cost effectiveness compared to the current gold standard treatment of parent + child. Results of these studies will be utilized as evidence to recommend changes in the standard treatment for childhood obesity. This program of research is critical for exploring and developing interventions that mobilize parents to intervene with their overweight and obese children. The timing of this research is optimal given the increase in childhood obesity in the United States, and the need for disseminative intervention and prevention programs.

ELIGIBILITY:
Inclusion Criteria:

* Overweight child 8-12 years of age and above the 95th% for age and gender
* An overweight (BMI > 25) parent willing to participate and attend all treatment meetings
* Eligible parent who can read at a minimum of an 8th grade level
* Family willing to commit to 5 months of treatment attendance, and follow-up for 18 months post-treatment.

Exclusion Criteria:

* Major child psychiatric disorder diagnoses
* Child diagnoses of a serious current physical disease (such as diabetes) for which physician supervision of diet and exercise prescription are needed (self-report)
* Family with restrictions on types of food, such as food allergies, religious, or ethnic practices that limit the foods available in the home
* Child with physical difficulties that limit the ability to exercise
* Child with an active eating disorder (based on EDE interview)
* Families where children or parents are involved in swimming or weight training more than 5 hours per week
* Major parent psychiatric disorder

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2010-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of parent-only treatment versus parent + child treatment on the body weight of the target child | At post-treatment visit (after 6-month treatment)
  The primary hypothesis is that the parent-only treatment will produce a decrease in the target child's weight (BMI for age percentile/BMI_Z) that is not inferior to the parent + child treatment immediately following treatment.
To evaluate the efficacy of parent-only treatment versus parent + child treatment on the body weight of the target child | At post-treatment 6-month follow-up visit
  The primary hypothesis is that the parent-only treatment will produce a decrease in the target child's weight (BMI for age percentile/BMI_Z) that is not inferior to the parent + child treatment at post-treatment 6-month follow-up visit.
To evaluate the efficacy of parent-only treatment versus parent + child treatment on the body weight of the target child | At post-treatment 18-month follow-up visit
  The primary hypothesis is that the parent-only treatment will produce a decrease in the target child's weight (BMI for age percentile/BMI_Z) that is not inferior to the parent + child treatment at post-treatment 18-month follow-up visit.

SECONDARY OUTCOMES:
To evaluate the cost-effectiveness of parent-only treatment versus parent + child treatment | At post-treatment visit (after 6-month treatment)
  We predict that the parent-only treatment will be more cost-effective than the parent + child group, as measured by calculating cost effectiveness ratios from both third party payer and limited societal perspectives at post-treatment visit (after 5-month treatment).
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's dietary quality | At post-treatment (after 6-month treatment)
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's dietary quality that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaire measures specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's exercise behavior | At post-treatment visit (after 6-month treatment)
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's exercise behavior that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's quality of life | At post-treatment visit (after 6-month treatment)
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's quality of life consisting of physical comfort, body esteem, social life, and family relations that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's psychosocial measures | At post-treatment visit (after 6-month treatment)
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's psychosocial measures, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on parent's adherence | At post-treatment visit (after 6-month treatment)
  We hypothesize that the parent-only treatment will produce an effect on the parent's adherence that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by group attendance and adherence to behavior recommendations.
To compare effect of parent-only treatment versus parent + child treatment on parenting style | At post-treatment visit (after 6-month treatment)
  We hypothesize that the parent-only treatment will produce an effect on the parenting style that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on parent's weight loss | At post-treatment visit (after 6-month treatment)
  We hypothesize that the parent-only treatment will produce parent weight loss (as measured by BMI) that is not inferior to the parent + child treatment.
To evaluate the predictors of success in childhood obesity treatments by evaluating change in target child's and parent's weight | At post-treatment visit (after 6-month treatment)
  A decrease in BMI percentile for age for target child and a decrease in BMI for parent will be evaluated.
To evaluate the predictors of success in childhood obesity treatments by evaluating compliance | At post-treatment visit (after 6-month treatment)
  Compliance will be measured by group attendance and adherence to behavior recommendations.
To evaluate the predictors of success in childhood obesity treatments by evaluating changes in household food environment | At post-treatment visit (after 6-month treatment)
  Changes in household food environment will be evaluated by assessing questionnaires specific for household food environment (Food Shelf Inventory).
To evaluate the predictors of success in childhood obesity treatment by evaluating change in parenting style | At post-treatment visit (after 6-month treatment)
  Changes in parenting style will be evaluated by assessing questionnaires that are specific to parenting style for child and parent.
To evaluate the predictors of success in childhood obesity treatment by evaluating changes in target child's and parent's psychosocial functioning | At post-treatment visit (after 6-month treatment)
  Changes in the target child's and parent's psychosocial functioning will be evaluated by assessing questionnaire measures specific to child and parent psychosocial functioning.
To evaluate the cost-effectiveness of parent-only treatment versus parent + child treatment | At post-treatment 6-month follow-up visit
  We predict that the parent-only treatment will be more cost-effective than the parent + child group, as measured by calculating cost effectiveness ratios from both third party payer and limited societal perspectives at post-treatment 6-month follow-up visit.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's dietary quality | At post-treatment 6-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's dietary quality that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaire measures specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's dietary quality | At post-treatment 18-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's dietary quality that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaire measures specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's exercise behavior | At post-treatment 6-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's exercise behavior that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's exercise behavior | At post-treatment 18-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's exercise behavior that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's quality of life | At post-treatment 6-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's quality of life consisting of physical comfort, body esteem, social life, and family relations that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's quality of life | At post-treatment 18-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's quality of life consisting of physical comfort, body esteem, social life, and family relations that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's psychosocial measures | At post-treatment 6-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's psychosocial measures, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on target child's and parent's psychosocial measures | A post-treatment 18-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the target child's and parent's psychosocial measures, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on parent's adherence | At post-treatment 6-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the parent's adherence that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by group attendance and adherence to behavior recommendations.
To compare effect of parent-only treatment versus parent + child treatment on parent's adherence | At post-treatment 18-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the parent's adherence that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by group attendance and adherence to behavior recommendations.
To compare effect of parent-only treatment versus parent + child treatment on parenting style | At post-treatment 6-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the parenting style that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on parenting style | At post-treatment 18-month follow-up visit
  We hypothesize that the parent-only treatment will produce an effect on the parenting style that will support weight loss, of which is not inferior to the parent + child treatment. The effect will be measured by assessing questionnaires specific for child and parent.
To compare effect of parent-only treatment versus parent + child treatment on parent's weight loss | At post-treatment 6-month follow-up visit
  We hypothesize that the parent-only treatment will produce parent weight loss (as measured by BMI) that is not inferior to the parent + child treatment.
To compare effect of parent-only treatment versus parent + child treatment on parent's weight loss | At post-treatment 18-month follow-up visit
  We hypothesize that the parent-only treatment will produce parent weight loss (as measured by BMI) that is not inferior to the parent + child treatment.
To evaluate the predictors of success in childhood obesity treatments by evaluating change in target child's and parent's weight | At post-treatment 6-month follow-up visit
  A decrease in BMI percentile for age for target child and a decrease in BMI for parent will be evaluated.
To evaluate the predictors of success in childhood obesity treatments by evaluating change in target child's and parent's weight | At post-treatment 18-month follow-up visit
  A decrease in BMI percentile for age for target child and a decrease in BMI for parent will be evaluated.
To evaluate the predictors of success in childhood obesity treatments by evaluating compliance | At post-treatment 6-month follow-up visit
  Compliance will be measured by group attendance and adherence to behavior recommendations.
To evaluate the predictors of success in childhood obesity treatments by evaluating compliance | At post-treatment 18-month follow-up visit
  Compliance will be measured by group attendance and adherence to behavior recommendations.
To evaluate the predictors of success in childhood obesity treatments by evaluating changes in household food environment | At post-treatment 6-month follow-up visit
  Changes in household food environment will be evaluated by assessing questionnaires specific for household food environment (Food Shelf Inventory).
To evaluate the predictors of success in childhood obesity treatments by evaluating changes in household food environment | At post-treatment 18-month follow-up visit
  Changes in household food environment will be evaluated by assessing questionnaires specific for household food environment (Food Shelf Inventory).
To evaluate the predictors of success in childhood obesity treatment by evaluating change in parenting style | At post-treatment 6-month follow-up visit
  Changes in parenting style will be evaluated by assessing questionnaires that are specific to parenting style for child and parent.
To evaluate the predictors of success in childhood obesity treatment by evaluating change in parenting style | At post-treatment 18-month follow-up visit
  Changes in parenting style will be evaluated by assessing questionnaires that are specific to parenting style for child and parent.
To evaluate the predictors of success in childhood obesity treatment by evaluating changes in target child's and parent's psychosocial functioning | At post-treatment 6-month follow-up visit
  Changes in the target child's and parent's psychosocial functioning will be evaluated by assessing questionnaire measures specific to child and parent psychosocial functioning.
To evaluate the predictors of success in childhood obesity treatment by evaluating changes in target child's and parent's psychosocial functioning | At post-treatment 18-month follow-up visit
  Changes in the target child's and parent's psychosocial functioning will be evaluated by assessing questionnaire measures specific to child and parent psychosocial functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, PhD, Principal Investigator — UCSD
Locations (1):
- UCSD Center for Healthy Eating and Activity Research (CHEAR), La Jolla, California, United States

REFERENCES:
- [Background] Bauer KW, Nelson MC, Boutelle KN, Neumark-Sztainer D. Parental influences on adolescents' physical activity and sedentary behavior: longitudinal findings from Project EAT-II. Int J Behav Nutr Phys Act. 2008 Feb 26;5:12. doi: 10.1186/1479-5868-5-12. PMID 18302765
- [Background] Epstein LH. Family-based behavioural intervention for obese children. Int J Obes Relat Metab Disord. 1996 Feb;20 Suppl 1:S14-21. PMID 8646260
- [Background] Epstein LH, Wing RR, Steranchak L, Dickson B, Michelson J. Comparison of family-based behavior modification and nutrition education for childhood obesity. J Pediatr Psychol. 1980 Mar;5(1):25-36. doi: 10.1093/jpepsy/5.1.25. No abstract available. PMID 7452420
- [Background] Epstein LH, Valoski A, Wing RR, McCurley J. Ten-year follow-up of behavioral, family-based treatment for obese children. JAMA. 1990 Nov 21;264(19):2519-23. PMID 2232019
- [Background] Wang G, Dietz WH. Economic burden of obesity in youths aged 6 to 17 years: 1979-1999. Pediatrics. 2002 May;109(5):E81-1. doi: 10.1542/peds.109.5.e81. PMID 11986487
- [Background] Birch LL, Davison KK. Family environmental factors influencing the developing behavioral controls of food intake and childhood overweight. Pediatr Clin North Am. 2001 Aug;48(4):893-907. doi: 10.1016/s0031-3955(05)70347-3. PMID 11494642
- [Background] Faith MS, Scanlon KS, Birch LL, Francis LA, Sherry B. Parent-child feeding strategies and their relationships to child eating and weight status. Obes Res. 2004 Nov;12(11):1711-22. doi: 10.1038/oby.2004.212. PMID 15601964
- [Background] Clark HR, Goyder E, Bissell P, Blank L, Peters J. How do parents' child-feeding behaviours influence child weight? Implications for childhood obesity policy. J Public Health (Oxf). 2007 Jun;29(2):132-41. doi: 10.1093/pubmed/fdm012. Epub 2007 Apr 18. PMID 17442696
- [Derived] Boutelle KN, Kang Sim DE, Eichen DM, Manzano MA, Rhee KE, Strong DR. Predictors of parent self-monitoring patterns in a family-based behavioral weight loss treatment program. Int J Obes (Lond). 2024 Oct;48(10):1457-1464. doi: 10.1038/s41366-024-01574-8. Epub 2024 Jul 15. PMID 39009764
- [Derived] Kang Sim DE, Strong DR, Manzano MA, Rhee KE, Boutelle KN. Evaluation of dyadic changes of parent-child weight loss patterns during a family-based behavioral treatment for obesity. Pediatr Obes. 2020 Jun;15(6):e12622. doi: 10.1111/ijpo.12622. Epub 2020 Feb 12. PMID 32048808
- [Derived] Eichen DM, Strong DR, Rhee KE, Rock CL, Crow SJ, Epstein LH, Wilfley DE, Boutelle KN. Change in eating disorder symptoms following pediatric obesity treatment. Int J Eat Disord. 2019 Mar;52(3):299-303. doi: 10.1002/eat.23015. Epub 2019 Jan 14. PMID 30638271
- [Derived] Boutelle KN, Rhee KE, Liang J, Braden A, Douglas J, Strong D, Rock CL, Wilfley DE, Epstein LH, Crow SJ. Effect of Attendance of the Child on Body Weight, Energy Intake, and Physical Activity in Childhood Obesity Treatment: A Randomized Clinical Trial. JAMA Pediatr. 2017 Jul 1;171(7):622-628. doi: 10.1001/jamapediatrics.2017.0651. PMID 28558104